CLINICAL TRIAL: NCT00306280
Title: Phase 1 Study of Phototherapy System to Treat H Pylori
Brief Title: Feasibility Study of Phototherapy System to Treat H Pylori
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LumeRx (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lmrx01
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Helicobacter Pylori
Keywords: Helicobacter pylori; phototherapy; peptic ulcer; gastric cancer
MeSH Terms: conditions — Peptic Ulcer; Stomach Neoplasms | interventions — Phototherapy

INTERVENTIONS:
Device: Phototherapy

SUMMARY:
This purpose of this study is to determine whether phototherapy can be used to safely and effectively treat H pylori.

DETAILED DESCRIPTION:
H pylori causes almost all peptic ulcers and many gastric cancers and is widely prevalent worldwide. Treatment by multiple antibiotics and proton pump inhibitors is effective but are compromised today by significant non compliance due to side effects and duration of required treatment. Also, the increase in antibiotic resistance coupled with the decreased availability of new antibiotics project a significant population of patients who will not be treatable with antibiotics.

A special, visible-light based phototherapy system has been demonstrated to significantly decrease the viability of H pylori in vitro and in a brief clinical experiment.

This study will evaluate the safety and short term efficacy in up to 60 patients of the phototherapy system to treat H pylori.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 90
* Documented positive for H. pylori infection by urease breath test, stool antigen or histology within thirty days prior to procedure
* Willing to comply with study requirements
* Able to undergo endoscopic esophagogastroduodenoscopy (EGD) with biopsy

Exclusion Criteria:

* History of gastric or duodenal carcinoma
* History of prior gastric or duodenal surgery
* Oral or intravenous antibiotics use within previous one month
* Use of bismuth subsalicylate (Pepto Bismol) within previous one month
* Use of photosensitizing drugs or nutritional supplements within previous one month
* Active peptic ulcer disease (gastric or duodenal ulcer)
* Esophagitis Grade II or higher
* Oral or intravenous antibiotics use within previous one month
* History of a bleeding disorder or anti-coagulant use that would prevent biopsy
* PPI treatment two weeks prior to the scheduled endoscopy
* Positive Pregnancy Test
* Known porphyria
* Suffer from phenylketonuria (PKU)
* Signs of jaundice
* Weight < 100 lb or > 250 lb
* Previously enrolled in this study
* Participating in another ongoing clinical trial in which concomitant diagnosis or therapeutic intervention would adversely affect the integrity of this study
* The subject is inappropriate for study participation, as determined by the Investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-03; Study Completion 2007-03

PRIMARY OUTCOMES:
Negative urease breath test at five weeks post procedure

SECONDARY OUTCOMES:
Procedural Side Effects
Negative urease breath test at 5 days post procedure
Reduction in acute post treatment bacterial population with respect to pretreatment samples

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Abbott Northwestern Hospital, Minneapolis, Minnesota